CLINICAL TRIAL: NCT02161055
Title: Randomized Controlled Clinical Study of Intensive Versus Nonintensive Insulin Therapy for Hyperglycemia After Traumatic Brain Injury
Brief Title: Intensive Versus Nonintensive Insulin Therapy for Hyperglycemia After Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lianyungang Oriental Hospital (Other)
Collaborators: The First People's Hospital of Lianyungang (Other)
Responsible Party: Principal Investigator, Wenxue Wang, Professor, Director of the Department of Neurosurgery, Lianyungang Oriental Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYG-1401-WW
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Brain Injuries; Hyperglycemia
Keywords: Insulin; Hyperglycemia; Postoperative Mortality; Intensive insulin therapy; Non-intensive insulin therapy; Brain Injuries; Wounds and Injuries; Craniocerebral Trauma; Trauma, Nervous System
MeSH Terms: conditions — Brain Injuries; Hyperglycemia; Insulin Resistance; Wounds and Injuries; Craniocerebral Trauma; Trauma, Nervous System | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Strict control group (Experimental): Intensive insulin therapy: Keep Target blood glucose levels between 4.4-7.0 mmol/L;
  Blood glucose levels were monitored and controlled using the Yale Insulin Infusion Protocol. Rapid blood glucose levels were monitored once every 2 hours.
  Interventions: Drug: Insulin
- Moderate control group (Experimental): Intensive insulin therapy: Keep target blood glucose levels between 7.1 and 10.0 mmol/L.
  Blood glucose levels were monitored and controlled using the Yale Insulin Infusion Protocol. Rapid blood glucose levels were monitored once every 2 hours
  Interventions: Drug: Insulin
- Slight control group (Experimental): Intensive insulin therapy: Keep target blood glucose levels between 10.1 and 13.0 mmol/L.
  Blood glucose levels were monitored and controlled using the Yale Insulin Infusion Protocol. Rapid blood glucose levels were monitored once every 2 hours.
  Interventions: Drug: Insulin
- Non-intensive insulin therapy (Active Comparator): Rapid blood glucose levels were measured once every 2 hours. When blood glucose levels were ≤ 13.0 mmol/L, no intervention was performed; When blood glucose levels were > 13.0 mmol/L, regular insulin was subcutaneously injected separately. During fasting, insulin was injected once every 8 hours. During venous or enteral nutrition infusion, insulin was infused at 30 minutes before nutrition infusion. When blood glucose levels were ≤ 13.0 mmol/L, insulin infusion was terminated.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin dose was selected in accordance with the Yale Insulin Infusion Protocol.
  • Amount of insulin (u) = [fasting blood glucose (mmol/L) × 18-100] × 10 × body weight (kilogram) × 0.6 ÷ 1000 ÷ 2
  Other Names: Insulin Injection(10mL:400u), manufactured by Wanbang Biochemical Pharmaceutical Co., Ltd. Lot No. 1307230, No. 1302225, No. 1307210.

SUMMARY:
An increase in blood glucose is a common clinical symptom in patients following traumatic brain injury. Studies confirm that death after traumatic brain injury was not only associated with nerve injury, but also correlated with abnormal physiological and metabolic reactions. Hyperglycemia is a manifestation of physiological and metabolic disorders after traumatic brain injury. Traumatic brain injury induced hyperglycemia, and then aggravated secondary injury to the brain. Therefore, it is of important clinical significance to study the treatment of hyperglycemia after traumatic brain injury.

DETAILED DESCRIPTION:
Hyperglycemia induced by traumatic brain injury is directly correlated with patient prognosis. Previous studies showed that if blood glucose could be controlled < 6.11 mmol/L, prognosis would be good and mortality would be decreased by approximately 50%. Moreover, the incidence of ICU-related complications, especially infection, was obviously reduced. A study concerning severe traumatic brain injury analyzed the recovery of patients at 18 days, 3 months and 1 year after trauma, and demonstrated that the prognosis of patients with blood glucose levels < 11.1 mmol/L within 24 hours of hospital admission was apparently better than those whose blood glucose levels were > 11.1 mmol/L. Hyperglycemia occurred after traumatic brain injury and was treated with intensive insulin therapy. Thus, blood glucose levels were controlled between 4.4 and 6.1 mmol/L, which noticeably shortened insulin use and decreased the incidence of multiple organ dysfunction and mortality of patients with traumatic brain injury.

It is well known that hyperglycemia will appear after traumatic brain injury. However, there are few clinical studies addressing continuous dynamic monitoring of blood glucose of traumatic brain injury patients and the relationship between changes in blood glucose and the degree of traumatic brain injury. Insulin therapy for reducing injury to secondary nerve cells after traumatic brain injury and for improving functional prognosis has also not been explored.

When blood glucose level is > 7.0 mmol/L as measured twice by rapid examination within 2 hours of hospital admission, patients with hyperglycemia after severe closed traumatic brain injury will be randomly divided into the intensive therapy group and nonintensive therapy group according to the random number table.

Patients in both groups will be treated using the protocol as follows.

1. Craniotomy for traumatic brain injury to mainly decompress and remove hematoma. Standard trauma craniotomy and incision of trachea will be performed.
2. During the operation, all patients will undergo ventricular puncture. Cerebrospinal fluid will be obtained for biochemical analysis and cell culture.
3. All patients will be closely monitored in the ICU of the Department of Neurosurgery.
4. Therapeutic protocols for severe traumatic brain injury will be used.
5. Glucocorticoid can cause disorders of glucose metabolism, so glucocorticoids can not be regularly applied in these two groups.
6. When glucose was injected into the vein, insulin was added at the proportion of 5:1 to eliminate glucose effects on blood glucose.

Blood glucose measurement: Capillary blood will be obtained from the tip of the ring finger to measure blood glucose. For a period, the blood should be collected from the same finger to make sure an accurate measurement occurs. When blood glucose of a patient undergoing transfusion was measured, blood should be collected from the tip of the finger of the limb without transfusion to ensure the accuracy of measurement.

Monitoring of target blood glucose: insulin dose will be selected in accordance with the Yale Insulin Infusion Protocol.

1. Insulin will be infused into the vein using a micropump at 0.1 μ/kg•h;
2. When blood glucose levels are > 20.0 mmol/L, insulin will be infused at 10.0 μ/h;
3. When blood glucose levels are between 17.1 and 20.0 mmol/L, insulin will be infused at 8.0 μ/h;
4. When blood glucose levels are between 14.1 and 17.0 mmol/L, insulin will be infused at 6.0 μ/h;
5. When blood glucose levels are between 11.5 and 14.0 mmol/L, insulin will be infused at 4.0 μ/h;
6. Within 12 and 24 hours, blood glucose levels will be maintained within the range of target blood glucose. During this period, blood glucose levels will be monitored once every 2 hours, and insulin dose will be adjusted in time.
7. If blood glucose levels are higher than the target value, insulin dose could be gradually increased by 1-2 μ/h;
8. When blood glucose levels reach the target value, insulin dose could be gradually diminished until terminated.

ELIGIBILITY:
Inclusion Criteria:

* Severe closed traumatic brain injury diagnosed in the clinic;
* Severe closed traumatic brain injury verified by CT examinations;
* Patients who are in accordance with the indications of craniotomy for severe traumatic brain injury;
* Blood glucose levels > 7.0 mmol/L measured twice by rapid examination within 2 hours of hospital admission;
* Glasgow coma score between 3 and 8;
* At the age of 18 - 80 years old;
* Irrespective of gender.

Exclusion Criteria:

* At the age of < 18 years old or > 80 years old;
* Glasgow coma score > 8;
* Patients combined with multiple site damage;
* Hemodialysis-dependent patients combined with diabetic nephropathy;
* Patients with nervous system disease before traumatic brain injury;
* Patients with a history of diabetes before suffering from a traumatic brain injury.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Monitoring of target blood glucose | 4 weeks
  Within 1 week of hospitalization, rapid blood glucose levels will be recorded once every 2 hours in each group. Glycosylated serum protein levels will be measured once a week, for 4 consecutive weeks. This index reflects the mean blood glucose levels of 2 - 3 weeks.

SECONDARY OUTCOMES:
Mortality | 6 months after surgery
  Percentage of patients who die during hospitalization period, at 1 week after surgery, at 2 weeks after surgery, and at 3 months after injury.
Evaluation of activity of daily living | 2 weeks after hospital admission, 3 months and 6 months after injury
  At 2 weeks after hospital admission, Modified Rankin Scale and Glasgow outcome score will be applied.
  During follow-up at 3 months after injury, Barthel index, Glasgow outcome score and Modified Rankin Scale will be employed.
  During follow-up at 6 months after injury, Barthel index and Glasgow outcome score will be used.

OTHER OUTCOMES:
Evaluation of severity of patient's condition | An expected time of 7 days
  Glasgow coma score will evaluate the severity of patient's condition, as will a recording sheet evaluating the patient's condition at hospital admission. Acute Physiology and Chronic Health Evaluation II will occur on each subsequent day in ICU.
CT monitoring of morphological changes in the brain | Until 14 days after surgery
  CT scans will monitor the morphological changes in the brain on hospital admission, preoperation, 1-3 days postoperation, 7 days postoperation, and 14 days postoperation.
Monitoring of changes in cerebrospinal fluid | 1 week after surgery
  Cerebrospinal fluid will be obtained for biochemical analysis and cell culture. Cerebrospinal fluid will be collected during surgery, and obtained at 1 week after surgery by lumbar puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxue Wang, M.D., Ph.D., Principal Investigator — Lianyungang Oriental Hospital
Locations (2):
- China (2):
  - Lianyungang Oriental Hospital, Lianyungang, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu

REFERENCES:
- [Derived] Yuan T, He H, Liu Y, Wang J, Kang X, Fu G, Xie F, Li A, Chen J, Wang W. Association between blood glucose levels and Glasgow Outcome Score in patients with traumatic brain injury: secondary analysis of a randomized trial. Trials. 2022 Jan 15;23(1):38. doi: 10.1186/s13063-022-06005-5. PMID 35033158